CLINICAL TRIAL: NCT04093544
Title: Expanding the Therapeutic Window of Deep Brain Stimulation in Parkinson's Disease by Means of Directional Leads: a Double-blind Cross-over Pilot Study
Brief Title: Expanding the Therapeutic Window of Deep Brain Stimulation in Parkinson's Disease by Means of Directional Leads
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Alfonso Fasano, Professor of Neurology, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 17-5705
Record Dates: First submitted 2019-09-07; First posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Parkinson Disease
Keywords: deep brain stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Stimulation (Active Comparator): Participants will receive stimulation using the best contact combination in ring mode.
  Interventions: Device: Deep brain stimulation
- Directional Stimulation (Experimental): Participants will receive stimulation using the best segmented (steered) contacts.
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Steered stimulation using directional leads

SUMMARY:
Exploring directional lead

DETAILED DESCRIPTION:
This is a single-centre, double-blinded cross-over study comparing the standard electrode configuration (ring-mode) vs. directional electrode configuration for steered stimulation of deep brain stimulation (DBS) patients.

The study will follow 2 phases.

Phase 1:

Visit 1 Screening/Baseline (T0):

As per current standard care for patients undergoing subthalamic deep brain stimulation (STN-DBS), participants will be screened 3-6 months before the DBS STN implant surgery (T0) according to the inclusion/exclusion criteria.

Visits for standard practiced care for programing of DBS Between 1 to 3 months after the surgery, programing of the DBS system for the 20 patients will be done in an open label fashion in order to find the contact able to reduce the motor symptoms without the side effects. This will be done according to the standard of practice currently adopted at Toronto Western Hospital.

Phase 2:

Visit 1

Randomization: 4 months +/- 4weeks after the surgery, patients will be randomized to two type of stimulation:

1. Standard : The percentage of current allocated to the central split contacts will be evenly distributed in order to perfectly mimic a standard ring contact. All possible types of frequencies and pulse widths will be used. The same amount of current for each of the active contacts will be used.
2. Directional: contacts 1-8 will be used in any possible configuration and using different amount of current for each of the active one as well as different frequencies. In conclusion, all the capabilities of the DBS system will be used.

Possible adjustments to stimulation parameters (e.g. pulse width, amplitude threshold) will be performed to achieve an optimal therapeutic window for each patient.

Visit 2 Follow up visit at 6 months +/- 4 weeks of the surgery for neurological examination if required.

Visit 3 (T1):

Cross over : 7 months +/- 4 weeks after the surgery patients will be switched to the other type of stimulation . Raters and patients will be blinded to the group allocation.

Visit 4:

Follow up visit at 9 months +/- 4 weeks of the surgery for neurological examination if required.

Visit 5 (T2):

End of study visit at month 10 +/- 4 weeks after the surgery. There might be unscheduled visits in case of unexpected clinical conditions (i.e. occurrence of side effects or worsening of motor conditions). Participants will be in this study for a maximum of 16 months. Throughout the whole study, participants will visit the clinic without their regular medication as part of standard treatment practice. All the stimulation adjustment will be performed by the same unblinded physician or sub-investigator.

ELIGIBILITY:
1. Patients with a diagnosis of Parkinson's disease (PD) according to the British Parkinson's Disease Society Brain Bank criteria, who fulfilled the inclusion and exclusion criteria proposed by the core assessment programme for surgical interventional therapies in PD panel
2. Male and female patients with idiopathic PD, who have symptoms responsive to L- dopa medications, but who have significant impairment related to PD that is no longer well controlled with pharmacotherapy (i.e., refractory to optimized medical therapy)
3. Patients considered as subthalamic nucleus deep brain stimulation (STN-DBS) candidates as per current standard of care. These patients will subsequently undergo STN-DBS surgery and maintain stimulation therapy.
4. Patients aged 18 to 80 years.
5. Quality of life and social functioning influenced by levodopa-responsive symptoms 6) No major comorbidities

Exclusion criteria will include patients with other significant neurologic or psychiatric illnesses or cognitive deficit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2020-05-15 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Number/incidence of adverse events | Throughout the study, averaging 6 months
  Number/incidence of adverse events

SECONDARY OUTCOMES:
Change from baseline in a measure of health related quality of life and non-motor symptoms of Parkinson's disease using the Parkinson's disease Questionnaire (PDQ-39) | After 3 months of each intervention
  The PDQ-39 assesses individuals experiences across 8 dimensions of daily living. Each dimension is scored from 0 to 100. Lower scores mean better quality of life.
Patients Global Impression of Change (PGIC) | After 3 months of each intervention
  The PGIC evaluates all aspects of patients' health and assesses if there has been an improvement or decline in clinical status relative to baseline. This is a seven point scale, lower values indicating worsening and higher values, improvement.
Change in articulation rate of speech using a Phonetics Software | After 3 months of each intervention
  Sample speeches will be recorded and digitalized at 44,000Hz using a microphone and analyzed with a Phonetics software. Articulation rate is calculated as the number of syllables produced/total time without pauses.
Change in dysfluency of speech using a Phonetics Software | After 3 months of each intervention
  Sample speeches will be recorded and digitalized at 44,000Hz using a microphone and analyzed ina Phonetics software. Dysfluency is calculated as percentage of dysfluent words/total number of words. Dysfluent words are defined as part-words, word or phrase repetitions, revisions, hesitations or fillers.
Change in intelligibility of speech using a Phonetics Software | After 3 months of each intervention
  Sample speeches will be recorded and digitalized at 44,000Hz using a microphone and analyzed in a Phonetics software. Intelligibility is a subjective measure of speech quality, and will be measured by a single rater trained in speech-language pathology.
Change in the Movement Disorders sponsored Unified Parkinson's disease Rating Scale (MDS-UPDRS), a measure of various motor and non-motor symptoms used to assess the clinical course of Parkinson's longitudinally. | After 3 months of each intervention
  The MDS-UPDRS scores range from 0 to 272, with higher scores meaning more severe disease
Change in the presence and severity of depressive symptoms using the Beck Depression Inventory (BDI) | After 3 months of each intervention
  The BDI is a 21-question multiple-choice self-report inventory for measuring the severity of depression. Scores range from 0 to 63, with higher scores meaning worse depression.
Walking speed measured with the Zeno Walkway | After 3 months of each intervention
  The Zeno Walkway is a 20 feet walking mat containing 16-pressure sensing pads and circuitry that allows for measurement of various gait and balance variables during straight walking. Patients will be asked to walk on the mat at a self selected pace. Walking speed will be measured.
Step length measured with the Zeno Walkway | After 3 months of each intervention
  The Zeno Walkway is a 20 feet walking mat containing 16-pressure sensing pads and circuitry that allows for measurement of various gait and balance variables during straight walking. Patients will be asked to walk on the mat at a self selected pace. Mean and coefficients of variation (standard deviation divided by the mean x 100) of step length will be measured.
Double support time measured with the Zeno Walkway | After 3 months of each intervention
  The Zeno Walkway is a 20 feet walking mat containing 16-pressure sensing pads and circuitry that allows for measurement of various gait and balance variables during straight walking. Patients will be asked to walk on the mat at a self selected pace. Mean and coefficients of variation (standard deviation divided by the mean x 100) of double support time will be measured. The double support time is the the time during gait where both feet are in contact to the ground
Cadence measured with the Zeno Walkway | After 3 months of each intervention
  The Zeno Walkway is a 20 feet walking mat containing 16-pressure sensing pads and circuitry that allows for measurement of various gait and balance variables during straight walking. Patients will be asked to walk on the mat at a self selected pace. Mean and coefficients of variation (standard deviation divided by the mean x 100) of cadence will be measured. Cadence is the number of steps per minute of walking.
Percentage of ON time without troublesome dyskinesias during waking hours | After 3 months of each intervention
  ON time without dyskinesias is defined as the period of time is which patients have good mobility, associated with a good response to treatments and without troublesome involuntary movements (dyskinesias). This will be measured as percentage of ON time during the waking hours of the day, Patients will complete 24-hours motor diaries during 3 consecutive days, in which they are asked to rate their motor functions every 30 minutes.
Number of falls or near-falls | Collected after 3 months of each intervention, but assessing all intervention period, averaging 6 months
  Participants will be asked to keep track of all falls and near-falls (an event in which a person feels a fall is imminent but avoids it by compensatory action, such as grabbing a nearby object or controlling the fall) on a written diary throughout the intervention period.
Change in levodopa equivalent daily dose (LEDD) | After 3 months of each intervention
  LEDD is calculated using a conversion formula to transform all medications used for treatment of Parkinson's disease to an equivalent dose of levodopa
Measure of resting-state local field potentials and functional connectivity of the brain using magnetoencephalography (MEG) | After 3 months of each intervention
  MEG will be used to measure the average absolute power and the power spectrum density of neuronal activity of the brain, both measures will be used to assess the effect of deep brain stimulation on the functional activity and oscillatory synchronization of various movement-related areas of the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Fasano, MD, Principal Investigator — University of Toronto
Locations (1):
- Movement disorders Centre, Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fasano A, Daniele A, Albanese A. Treatment of motor and non-motor features of Parkinson's disease with deep brain stimulation. Lancet Neurol. 2012 May;11(5):429-42. doi: 10.1016/S1474-4422(12)70049-2. PMID 22516078
- [Background] Herzog J, Pinsker M, Wasner M, Steigerwald F, Wailke S, Deuschl G, Volkmann J. Stimulation of subthalamic fibre tracts reduces dyskinesias in STN-DBS. Mov Disord. 2007 Apr 15;22(5):679-84. doi: 10.1002/mds.21387. PMID 17266046
- [Background] Barbe MT, Maarouf M, Alesch F, Timmermann L. Multiple source current steering--a novel deep brain stimulation concept for customized programming in a Parkinson's disease patient. Parkinsonism Relat Disord. 2014 Apr;20(4):471-3. doi: 10.1016/j.parkreldis.2013.07.021. Epub 2013 Sep 14. No abstract available. PMID 24041939
- [Background] Timmermann L, Jain R, Chen L, Maarouf M, Barbe MT, Allert N, Brucke T, Kaiser I, Beirer S, Sejio F, Suarez E, Lozano B, Haegelen C, Verin M, Porta M, Servello D, Gill S, Whone A, Van Dyck N, Alesch F. Multiple-source current steering in subthalamic nucleus deep brain stimulation for Parkinson's disease (the VANTAGE study): a non-randomised, prospective, multicentre, open-label study. Lancet Neurol. 2015 Jul;14(7):693-701. doi: 10.1016/S1474-4422(15)00087-3. Epub 2015 May 28. PMID 26027940
- [Background] Contarino MF, Bour LJ, Verhagen R, Lourens MA, de Bie RM, van den Munckhof P, Schuurman PR. Directional steering: A novel approach to deep brain stimulation. Neurology. 2014 Sep 23;83(13):1163-9. doi: 10.1212/WNL.0000000000000823. Epub 2014 Aug 22. PMID 25150285
- [Background] Steigerwald F, Muller L, Johannes S, Matthies C, Volkmann J. Directional deep brain stimulation of the subthalamic nucleus: A pilot study using a novel neurostimulation device. Mov Disord. 2016 Aug;31(8):1240-3. doi: 10.1002/mds.26669. Epub 2016 May 31. PMID 27241197
- [Background] Pollo C, Kaelin-Lang A, Oertel MF, Stieglitz L, Taub E, Fuhr P, Lozano AM, Raabe A, Schupbach M. Directional deep brain stimulation: an intraoperative double-blind pilot study. Brain. 2014 Jul;137(Pt 7):2015-26. doi: 10.1093/brain/awu102. Epub 2014 May 19. PMID 24844728